CLINICAL TRIAL: NCT02866890
Title: The New Laryngeal Tube Suction-Disposable for Childrens. An Observational Study
Brief Title: The New Laryngeal Tube Suction-Disposable for Childrens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, M.D., Bnai Zion Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BnaiZionMC-16-LG-003
Record Dates: First submitted 2016-07-25; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Adverse Anesthesia Outcome
Keywords: Laryngeal Tube Suction; seal pressure; mechanical ventilation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Laryngeal Tube Suction size 1 (Experimental): Measurement of leak pressure
  Interventions: Device: Laryngeal Tube Suction
- Laryngeal Tube Suction size 2 (Experimental): Measurement of leak pressure
  Interventions: Device: Laryngeal Tube Suction
- Laryngeal Tube Suction size 2.5 (Experimental): Measurement of leak pressure
  Interventions: Device: Laryngeal Tube Suction

INTERVENTIONS:
Device: Laryngeal Tube Suction — Laryngeal Tube Suction Measurement of leak pressure
  Other Names: VBM Medical, Sulz, Germany

SUMMARY:
The Laryngeal Tube Suction Disposable( LTS-D) has recently undergone considerable structural changes in design. As these changes may influence the performance of the LTS-D relative to the old LTS-D version the investigator decided to check the new LTS-D in the pediatric version The investigator hypothesized that the LTS-D perform clinically well during general anesthesia with controlled ventilation.

DETAILED DESCRIPTION:
The LTS-D, is a second generation supraglottic airway device, made from the medical polyvinyl chloride introduce in 2005. It is used for maintaining the airway during spontaneous and controlled ventilation during general anesthesia . It has been advocated for prehospital emergency airway management and serves as a useful tool during failed intubations The LTS-D has recently undergone considerable changes in design based on clinical studies and investigators feedback. The new LTS-D is available to adult and pediatric sizes.For childrens the devices is presented in the size 3 for patients of < 155 cm (> 30 Kg.), the size 2.5 for patients 125-150cm. (20-30 Kg.), the size 2 for patients of 12-25 Kg, the size 1 for patients of 5-12 Kg and the size 0 for patients < 5 Kg.

As these changes may influence the performance of the LTS-D relative to the old LTS-D version the investigator decided to check the new LTS-D in the pediatric version.

The investigator hypothesized that the LTS-D perform clinically well during general anesthesia with controlled ventilation.

ELIGIBILITY:
Inclusion Criteria:Pediatric patients, ASA I and II, normal airway, for minor elective surgery

Exclusion Criteria: Weigth <10Kg or > 30 Kg, known difficult airway, active esophagial reflux

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Seal pressure in cm H2O | one minute
  We will measure the seal leak pressure at 60 cm H2O intracuff pressure and the minimal pressure of the cuff to performed effective volume controlled ventilation

SECONDARY OUTCOMES:
Time of insertion in seconds | one minute
  Was measured as the time after the anesthesiologist removed the facemask until the square-wave capnograph tracing was observed after insertion of the LTS-D. Two attempts at insertion were permitted.

OTHER OUTCOMES:
Easy of insertion using a five-point Likert Scale | One minute
  Investigators were asked to complete a questionnaire independently and anonymously to record the 'ease-of-use' of the LTS-D. Insertion of the devices was classified as 1= easy, 2= moderate, 3= difficult and 4=impossible.

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Gaitini, M.D., Principal Investigator — Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: Yes